CLINICAL TRIAL: NCT00217256
Title: A Randomized Controlled Trial of the Medtronic Endeavor Drug (ABT-578) Eluting Coronary Stent System Versus the Cypher Sirolimus-Eluting Coronary Stent System in De Novo Native Coronary Artery Lesions
Brief Title: The Medtronic Endeavor III Drug Eluting Coronary Stent System Clinical Trial
Acronym: ENDEAVOR III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: K. Bogdanovich, Medtronic Cardiovascular
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IP056
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Artery Disease
Keywords: Restenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Endeavor Drug Eluting Stent
  Interventions: Device: Percutaneous Coronary Stenting
- 2 (Active Comparator): Cypher Drug Eluting Stent
  Interventions: Device: Percutaneous Coronary Stenting

INTERVENTIONS:
Device: Percutaneous Coronary Stenting — Endeavor Drug Eluting Stent
  Arms: 1
Device: Percutaneous Coronary Stenting — Cypher Drug Eluting Stent
  Arms: 2

SUMMARY:
To demonstrate the equivalency in in-segment late lumen loss at 8 months between the Endeavor Drug Eluting Coronary Stent System coated with ABT-578 (10 micrograms/mm) and the Cypher Sirolimus-Eluting Coronary Stent System for the treatment of single de novo lesions in native coronary arteries 2.5-3.5 mm in diameter.

DETAILED DESCRIPTION:
The ENDEAVOR III Trial is a prospective, multi-center, single-blind, randomized trial that enrolled 436 patients at 29 sites in the US. The purpose of this trial is to demonstrate the equivalency of in-segment late lumen loss at 8 months between the Endeavor stent and the Cypher stent for the treatment of single de novo lesions in native coronary arteries 2.5-3.5 mm in diameter. Patients were randomized to receive the Endeavor stent or the Cypher Sirolimus-Eluting Coronary Stent System. Enrollment was completed in September 2004.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is at least 18 years of age.
2. The patient must have clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia, or a positive functional study.
3. The patient is an acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting, and emergent coronary artery bypass graft (CABG) surgery.
4. Female patients of childbearing potential must have a negative pregnancy test within seven (7) days before the procedure.
5. The patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board of the respective clinical site.
6. The patient and the treating physician agree that the patient will return to the treating research center, or an affiliated institution under the same IRB jurisdiction, for all required post-procedure follow-up visits. A research staff member who has been properly trained to the Endeavor III protocol must conduct all follow-up evaluations.

Exclusion Criteria:

1. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, cobalt, nickel, chromium, molybdenum, or a sensitivity to contrast media, which cannot be adequately pre-medicated.
2. History of an allergic reaction or significant sensitivity to drugs similar to ABT-578 (rapamycin or rapamycin analog).
3. A platelet count < 100,000 cells/mm³ or > 700,000 cells/mm³, or a WBC < 3,000 cells/mm³.
4. A creatinine level > 2.0 mg/dL.
5. Evidence of an acute myocardial infarction within 72 hours of the intended treatment (defined as: Q wave or non-Q wave myocardial infarction having creatine kinase (CK) enzymes greater than or equal to 2X the upper laboratory normal with the presence of a creatine kinase myocardial-band isoenzyme (CK-MB) elevated above the Institution's upper limit of normal).
6. Any previous or planned treatment of any vessel with a drug eluting stent.
7. Previous or planned percutaneous coronary intervention of any vessel within 30 days pre or post procedure.
8. Previous stenting anywhere in the target vessel.
9. During the index procedure, the target lesion requires treatment with a device other than PTCA prior to stent placement (such as, but not limited to, cutting balloon, directional coronary atherectomy, excimer laser, rotational atherectomy, thrombectomy, etc.).
10. History of a stroke or transient ischemic attack within the prior 6 months.
11. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months.
12. History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
13. Concurrent medical condition with a life expectancy of less than 12 months.
14. Any previous or planned treatment of the target vessel with anti-restenotic therapies including, but not limited to brachytherapy.
15. Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints; or requires coronary angiography, intravascular ultrasound (IVUS) or other coronary artery imaging procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2004-02; Primary Completion 2005-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
In-segment late lumen loss | 8 months

SECONDARY OUTCOMES:
Device Success | 9 months
Lesion Success | 9 months
Procedure Success | 9 months
Major Adverse Cardiac Event (MACE) rate | 30 days, 6, 9, and 12 months
Target Site Revascularization (TSR) rate and clinically-driven TSR rate | 9 months
Target Vessel Revascularization (TVR) rate and clinically-driven TVR rate | 9 months
Target Vessel Failure (TVF) rate | 9 months
Angiographic binary restenosis (> 50% diameter stenosis) rate | 8 months
In-stent and in-segment minimum lumen diameter (MLD) | 8 months
Neointimal hyperplastic volume as measured by IVUS | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin B. Leon, M.D., Principal Investigator — Columbia University College of Physicians & Surgeons

REFERENCES:
- [Derived] Kandzari DE, Mauri L, Popma JJ, Turco MA, Gurbel PA, Fitzgerald PJ, Leon MB. Late-term clinical outcomes with zotarolimus- and sirolimus-eluting stents. 5-year follow-up of the ENDEAVOR III (A Randomized Controlled Trial of the Medtronic Endeavor Drug [ABT-578] Eluting Coronary Stent System Versus the Cypher Sirolimus-Eluting Coronary Stent System in De Novo Native Coronary Artery Lesions). JACC Cardiovasc Interv. 2011 May;4(5):543-50. doi: 10.1016/j.jcin.2010.12.014. PMID 21596327
- [Derived] Remak E, Manson S, Hutton J, Brasseur P, Olivier E, Gershlick A. Cost-effectiveness of the Endeavor stent in de novo native coronary artery lesions updated with contemporary data. EuroIntervention. 2010 Feb;5(7):826-32. doi: 10.4244/eijv5i7a138. PMID 20142198
- [Derived] Eisenstein EL, Leon MB, Kandzari DE, Mauri L, Edwards R, Kong DF, Cowper PA, Anstrom KJ; ENDEAVOR III Investigators. Long-term clinical and economic analysis of the Endeavor zotarolimus-eluting stent versus the cypher sirolimus-eluting stent: 3-year results from the ENDEAVOR III trial (Randomized Controlled Trial of the Medtronic Endeavor Drug [ABT-578] Eluting Coronary Stent System Versus the Cypher Sirolimus-Eluting Coronary Stent System in De Novo Native Coronary Artery Lesions). JACC Cardiovasc Interv. 2009 Dec;2(12):1199-207. doi: 10.1016/j.jcin.2009.10.009. PMID 20129546